CLINICAL TRIAL: NCT06889311
Title: Evaluation of Subperiosteal Hyaluronic Acid Injection Overlay Technique Compared to Tunneling with Connective Tissue Graft in Management of Interdental Papillary Defects: a Randomized Clinical Trial
Brief Title: A Modern, Non-surgical Method for Treating Papillary Deficiencies is the Use of Hyaluronic Acid, Which Have Demonstrated Encouraging Outcome. Subperiosteal Hyaluronic Acid Injection Overlay Technique with the Idea of Merging Hyaluronic Acid Injection with Surgical Intervention to Reconstruct Idp
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Amagad, Professor of Oral Medicine and Periodontology Faculty of Dentistry, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2024-12-16
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Interdental Papillae Reconstruction; Hyaluronic Acid
Keywords: Hyaluronic acid, Interdental papilla, Black triangle

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental)
  Interventions: Procedure: Subperiosteal hyaluronic acid injection overlay technique
- Group B (Active Comparator)
  Interventions: Procedure: Tunneling with connective tissue graft.

INTERVENTIONS:
Procedure: Subperiosteal hyaluronic acid injection overlay technique — using subperiosteal hyaluronic acid injection overlay technique showed promising results in treating lost interdental papilla which needs further assessment to its clinical effectiveness
  Arms: Group A
Procedure: Tunneling with connective tissue graft. — Connective tissue graft base techniques have been for years the most predictable approach for treatment of interdental papillary defects. CTG can as a biological filler which enhances flap stability and wound strength. CTG also can promote coagulation cascade and protects the maturating fibrin clot (Tavelli et al. 2019). Moreover, CTG results in significant increase in gingival tissue thickness which positively improve tissue fill and soft tissue volume creeping which influence esthetic outcomes following periodontal regeneration
  Arms: Group B

SUMMARY:
The interdental papilla is a crucial part of an esthetic smile, its loss results in gingival black triangles giving unpleasant appearance which directly affect patient self-esteem (Lee et al. 2016). The presence of interdental papilla is of great concern for the clinician and the patient. Gingival black triangles are considered to be the most disliked esthetic issue. As well open embrasures can cause food impaction and phonetic problems (Prato et al. 2004).

The treatment of black triangles is challenging in modern dentistry. The treatment options are surgical and non-surgical. Surgical treatments are invasive and do not always give a predictable result due to limited blood supply of the papilla (Mansouri 2013).

However, no technique has been set up as a gold standard treatment for gingival black triangles, although, connective tissue graft surgical techniques are the most common used approaches for treatment of black triangles (RahimiRad 2018).

A modern, non-surgical method for treating papillary deficiencies is the use of hyaluronic acid, which have demonstrated encouraging outcome (Ni et al. 2021). Subperiosteal hyaluronic acid injection overlay technique was proposed by Spano et al, (2020) with the idea of merging hyaluronic acid injection with simple surgical intervention to reconstruct the lost interdental papilla. As far as we know, there is no present studies comparing hyaluronic acid overlay technique with connective tissue graft in treatment of interdental papilla deficiencies.

DETAILED DESCRIPTION:
The interdental papilla is an important anatomical part of the gingiva. It can reduce by time or by different etiological factors as crown shape or presence of periodontal diseases which results in presence of highly unaesthetic black triangles which frequently cause patients complaints in both appearance and function (Patel et al. 2024). The interdental papilla is a part of the gingiva that fills the embrasure space between the contact point of the adjacent teeth. It is supported by the underlying alveolar bone and laterally by the presence of the teeth. It is composed of masticatory mucosa and composed of dense connective tissue covered with oral epithelium (Prato et al. 2004).

Tarnow et al (1992) investigated a relationship between the distance of interdental bone level and contact point and the presence or absence of the interdental papilla. They found that a distance of 3-4 mm, an intact interdental papilla was present. While, when the distance increased to 6 mm and above, there was partial or complete absence of the interdental papilla and the absence of the papilla increased with every millimeter. The interdental papilla can be lost due to interproximal bone loss due to periodontitis or may be iatrogenic damage such as over-countered restorations and crown preparations. In addition, tooth-related factors can cause loss of interdental papilla as loss of contact point, tooth malposition, abnormal tooth shape, triangular-shaped crowns, diastamas, divergent roots and over-eruption of a tooth (Kurth and Kokich 2001).

Nordland and Tarnow (1998) proposed a classification for the loss of interdental papilla which is based on three references: the contact point, buccal apical extent of the cemento-enamel junction (CEJ) and the interproximal CEJ. The classification follows: Normal: when the interdental papilla fills the embrasure space to contact point, Class I: the tip of the papilla lies between the interdental contact point and the most coronal extent of CEJ, Class II: the tip of the papilla lies at or apical to the interdental CEJ but coronal to facial CEJ and Class III: when the tip of the papilla lies at a level apical to the facial CEJ.

Different surgical and non-surgical techniques have been proposed for treatment of interdental papillary deficiency based on the etiological factor with some of degree of success. Among these treatments are the correction of traumatic oral hygiene practices, papilla enhancement with either autologous fibroblast injection or hyaluronic acid and orthodontic therapy (Singh et al. 2013). Among surgical approaches to reconstruct the lost papilla are connective tissue graft base surgical techniques. The surgical treatment of deficient papilla with the connective tissue graft remained the most used approach however, it requires a good vascular supply in the interdental papilla and requires a second surgical site (Gobbato et al. 2016).

Hyaluronic acid injection in the deficient interdental papilla has shown promising results (Fakhari and Berkland 2013; Lee et al. 2016; Ni et al. 2021). Hyaluronic acid is a polysaccharide present in the body tissues. Under physiologic conditions it binds to water and swells in a gel form, resulting in smoother tissue counters. The role of hyaluronic acid in augmentation is by inducing water absorption of gingival fibroblast proliferation. When hyaluronic acid is incorporated into an aqueous solution, hydrogen bonding occurs between adjacent carboxyl and N-acetyl groups; this feature allows hyaluronic acid to maintain conformational stiffness to retain water (Bertl et al. 2017). Also, it may affection collagen remodeling by increasing the production of procollagens and matrix metalloproteinase-1 secretion by fibroblast (Singh et al. 2013). Hyaluronic acid showed a satisfactory result in regeneration of lost interdental papilla at 6 and 12 months (Ficho et al. 2021).

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients aged over 18 years. 2. Class I papillary recession according to the Nordland and Tarnow classification system. (Nordland and Tarnow 1998) 3. Patients free from any systemic conditions that may affect healing. (Hamadeh et al. 2024).

4. The distance between the contact point to alveolar crest between 5 to 7 mm. 5. Presence of the adjacent teeth. 6. Compliant patients with good oral hygiene.

Exclusion Criteria:

- 1. Smokers. 2. Pregnant females. 3. Patients with active periodontal disease. 4. Patients who has spacing or crowding between the teeth to be treated. 5. Abnormal tooth shape or adjacent teeth with caries. 6. Presence of proximal restoration or orthodontic appliances or fixed prosthesis.

7. Patients with poor oral hygiene according to plaque index score of 2.0 to 3.0 evaluated according to the criteria of Silness and Loe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Changes in papilla height | Changes will be recorded at 3, 6 and 12 months
  Clinical changes in papilla will be recorded by measuring papilla height at the distance between the tip of the papilla and the incisal edge of the adjacent tooth using UNC periodontal probe .

SECONDARY OUTCOMES:
Percentage of changes in papilla height | 3, 6 and 12 months
  the percentage of change in papilla height will be calculated with a reference to baseline following equation PH baseline- PH timepoint / PH baseline
Papilla presence index | 3, 6 and 12 months
  The papilla presence index will be recorded at baseline, 3, 6 and 12 months follow up. The scores will be measured as follows: PPI 1: When the papilla is completely present and coronally extends to the contact point to completely fill the embrasure. It is at same level of adjacent papilla PPI 2: Papilla is no longer completely present and lies apical to the contact point and not at the same level as the adjacent papillae, but the interproximal CEJ is still not visible. PPI 3: Papilla is moved more apical and the interproximal CEJ becomes visible. PPI 4: Papilla lies apical to both the interproximal CEJ and buccal CEJ.
Clinical attachment loss | 3, 6 and 12 months
  A UNC probe will used to estimate this measurement. The probe will be inserted in the gingival sulcus and CAL will be measured as the distance from CEJ to the bottom of the sulcus
Gingival thickness | 3, 6 and 12 months
  Gingival thickness will be measured 2 mm apical to the gingival margin with an aesthetic needle with a silicon stopper. The needle will be inserted perpendicular to the mucosal surface, through soft tissue with light pressure until resistance will be felt once the tip of needle is in contact with bone. The silicone stopper will be moved towards until it reaches the external surface of mucosal tissues. The penetration depth will be measured using UNC graduated probe by measuring the distance from the tip of the needle to silicone stopper
Post-operative pain | 1,3 and 10 days post-surgical.
  Visual analogue scale (VAS) will be used to record post-operative pain. The pain will be measured as follows from 0, no pain to 10, maximum pain and will be measured at day 1,3 and 10 days post-surgical.
Patients' esthetic satisfaction | 12 months
  VAS will be used to record patients' esthetic satisfaction at six months. The satisfaction will be measured as follows (equal, better or worse than pre-surgery). Questionnaire will be taken for esthetic satisfaction, tooth brushing ability and dental hypersensitivity.
The need for analgesics | 10 days
  The pain will be measured indirectly by the total number of analgesic tablets that will be consumed by the patients after surgery by 10 days.

IPD SHARING:
Plan to Share IPD: Undecided